CLINICAL TRIAL: NCT00022230
Title: Combination of Chemotherapy With Taxol, Adriamycin, and Cytoxan (TAC), Multiple Infusions of Activated T Cells (ATC), Interleukin-2 (IL-2) and GM-CSF for High Risk Breast Cancer With and Without Her2/Neu Overexpression. (Phase I/II)
Brief Title: Combination Chemotherapy Plus Biological Therapy in Treating Patients With Stage II or Stage III Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left Institution
Sponsor: Roger Williams Medical Center (Other)
Responsible Party: Lawrence Lum, Roger Williams Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068797; RWMC-0633846
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — aldesleukin; Filgrastim; sargramostim; Cyclophosphamide; Doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin
Biological: filgrastim
Biological: sargramostim
Biological: therapeutic autologous lymphocytes
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies use different ways to stimulate the immune system and stop tumor cells from growing. Combining chemotherapy with biological therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects of giving chemotherapy together with biological therapy and to see how well they work in treating patients with stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects of sequential paclitaxel (or other taxane), doxorubicin, and cyclophosphamide followed by immunotherapy with activated T cells, interleukin-2, and sargramostim (GM-CSF) in patients with high-risk stage II or III breast cancer.
* Determine the disease-free survival and overall survival of patients treated with this regimen.
* Determine the immune function of patients treated with this regimen.

OUTLINE: Patients are stratified according to number of positive lymph nodes (less than 4 nodes vs 4-9 nodes vs 10 or more nodes), type of taxane chemotherapy during study (paclitaxel vs other taxane), and prior treatment with 2 of 3 study chemotherapy agents (yes vs no).

Patients receive doxorubicin IV on day 1 and filgrastim (G-CSF) on days 3-10 of 3 consecutive 14-day courses. Patients then receive paclitaxel or another taxane IV on day 1 and G-CSF on days 3-10 of 3 consecutive 14-day courses. Patients then receive cyclophosphamide IV on day 1 and G-CSF on days 3-10 of 3 consecutive 14-day courses. Patients who enroll after previously receiving 2 of these 3 chemotherapy drugs may receive the third. Treatment continues in the absence of disease progression or unacceptable toxicity.

After recovery from chemotherapy, patients undergo peripheral blood mononuclear cell (PBMC) collection. The PBMC are treated ex vivo with monoclonal antibody OKT3 to form activated T cells (ATC). The ATC are expanded for up to 14 days in interleukin-2 (IL-2).

At 3-4 weeks after PBMC collection, patients receive ATC IV over 15-30 minutes weekly for 8 weeks. Patients also receive IL-2 subcutaneously (SC) daily and sargramostim (GM-CSF) SC twice weekly beginning 3 days before the first ATC infusion and continuing until 7 days after completion of ATC therapy.

Patients are followed every 3 months for 1 year and then annually thereafter.

PROJECTED ACCRUAL: A total of 40-60 patients will be accrued for this study within 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage II or III adenocarcinoma of the breast
* High-risk disease

  * At least 4 positive lymph nodes
  * Fewer than 4 positive lymph nodes considered high-risk if one of the following is present:

    * HER2/neu-positive disease
    * Enlarged axillary nodes
    * Extra capsular extension of tumor from lymph node
    * Dermal lymphatic invasion
    * Vascular invasion
    * Bilateral disease
    * Familial breast cancer
    * T4 locally advanced disease
* Clinically chemosensitive to prior paclitaxel (or other taxane), doxorubicin, and cyclophosphamide

  * No relapse after chemotherapy
* No clinical evidence of brain metastases
* Hormone receptor status:

  * Estrogen and progesterone receptor status known

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100% OR
* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 50,000/mm^3
* Hemoglobin greater than 8 g/dL

Hepatic:

* Bilirubin less than 1.5 times normal
* SGOT less than 1.5 times normal

Renal

* Creatinine less than 1.8 mg/dL
* Creatinine clearance at least 60 mL/min
* BUN less than 1.5 times normal

Cardiovascular:

* Ejection fraction at least 45% by MUGA
* No uncontrolled or significant cardiovascular disease
* No myocardial infarction within the past year
* No significant congestive heart failure

Pulmonary:

* FEV_1 at least 60% predicted
* DLCO at least 60% predicted
* FVC at least 60% predicted

Other:

* No other malignancy except curatively treated squamous cell carcinoma in situ of the cervix or basal cell skin cancer
* No other serious medical or psychiatric illness that would preclude study participation
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* Prior standard chemotherapy with anthracyclines or combination chemotherapy involving a combination of taxanes, doxorubicin, and/or cyclophosphamide allowed

Endocrine therapy:

* No concurrent hormonal therapy for breast cancer
* Concurrent hormonal therapy for nondisease-related conditions (e.g., insulin for diabetes) allowed
* Concurrent steroids for adrenal failure, septic shock, or pulmonary toxicity allowed

Radiotherapy:

* Not specified

Surgery:

* Prior complete resection of tumor allowed

Other:

* Prior successful neoadjuvant therapy allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-01; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Toxicity
Disease-free survival
Overall survival
Immune functions

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence G. Lum, MD, DSc, Study Chair — Roger Williams Medical Center
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States